CLINICAL TRIAL: NCT01954329
Title: Markers in the Diagnosis of TIA
Acronym: MIND-TIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Saltro, diagnostic center for primary care. (Unknown)
Responsible Party: Principal Investigator, F.H. Rutten, MD, PhD, UMC Utrecht
Other Study IDs: NL43627.041.13
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Transient Ischemic Attack
Keywords: Biomarkers; TIA; Diagnosis
MeSH Terms: conditions — Ischemic Attack, Transient; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, RNA and DNA material.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients suspected of TIA by the GP

SUMMARY:
MIND-TIA is primarily an observational diagnostic study that aims to evaluate the role of novel biomarkers in the diagnosis of Transient Ischemic Attack (TIA)in primary care.

Rapid and adequate diagnosis of TIA is of great importance to enable a rapid start of treatment, and thereby decrease the risk of subsequent ischemic stroke.

DETAILED DESCRIPTION:
Rationale:

A Transient Ischaemic Attack (TIA) does not cause permanent damage of brain tissue, but the risk of a subsequent ischemic stroke in the short term is high. Timely recognition of TIA would result in early treatment and reduce the risk of ischaemic stroke, and other adverse cardiovascular events.

To improve the management of TIA adequate diagnosis is of imminent importance. However the diagnosis is notoriously difficult, for both GP and neurologist.

Adequate biomarkers for brain ischaemia could improve the early diagnosis and thus the subsequent management of TIA.

Objectives:

1. To assess the added diagnostic value of biomarkers beyond the clinical assessment (medical history, signs and symptoms) in patients suspected of TIA.

   Secondary objectives
2. To assess the prognostic value of biomarkers in patients with an established diagnosis of TIA.
3. To assess the time delay and factors related to delay in patients suspected of TIA.

Study population:

350 adult persons suspected of TIA from primary care.

Methods:

Recruitment of patients will be performed at the general practices of 200 GPs in the vicinity of 4 to 5 participating hospitals. During a home visit a research nurse collects a blood sample, and takes two health-related questionnaires. Participants will be referred by their GP to the regional TIA outpatient clinic for additional investigations, including brain imaging. The diagnostic accuracy of a set of biomarkers will be assessed with the 'definite' diagnosis of TIA by a panel of neurologists as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Being adult (18 years and older)
* Presenting to the GP with a new episode of symptoms suspected of TIA and the GP considering further investigations to confirm or exclude TIA at the TIA outpatient clinic.
* A blood sample can be collected within 72 hours after onset of symptoms.

Exclusion Criteria:

* The patient still has active symptoms or signs suspected of an ongoing ischemic stroke and immediate referral to the neurologist seems indicated.
* Valid history taking is impossible because of severe cognitive impairment or insufficient knowledge of the Dutch language.
* Patient with a life expectancy of < 6 months.
* Patient is not willing or able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 350 patients suspected of TIA by the GP
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
'Definite' Diagnosis of TIA | After 6 months of follow-up
  Determined by expert panel consisting of 3 neurologists

SECONDARY OUTCOMES:
Ischemic stroke and other cardiovascular events | During 6 months of follow-up
  Assessed in the medical records of the GPs
Time delay to GP consultation and start of treatment | 1 day of home visit

CONTACTS AND LOCATIONS:
Locations (1):
- Julius Center UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Dolmans LS, Rutten F, Bartelink MEL, van Dijk EJ, Nederkoorn PJ, Kappelle J, Hoes AW; MIND-TIA study group. Serum biomarkers in patients suspected of transient ischaemic attack in primary care: a diagnostic accuracy study. BMJ Open. 2019 Oct 17;9(10):e031774. doi: 10.1136/bmjopen-2019-031774. PMID 31628130
- [Derived] Dolmans LS, Rutten FH, El Bartelink ML, Seppenwoolde G, van Delft S, Kappelle LJ, Hoes AW. Serum biomarkers for the early diagnosis of TIA: The MIND-TIA study protocol. BMC Neurol. 2015 Jul 28;15:119. doi: 10.1186/s12883-015-0388-z. PMID 26215720
- See also: Dutch study website — http://www.juliuscentrum.nl/MIND-TIA